CLINICAL TRIAL: NCT06746428
Title: ACTIVATE: A Pilot Randomized Activity Coaching Trial to Increase Vitality and Energy During Post-operative Pelvic Radiation Therapy for Endometrial Cancer
Brief Title: Activity Coaching During Pelvic Radiation Therapy
Acronym: ACTIVATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inova Health Care Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INOVA-2024-91
Record Dates: First submitted 2024-12-17; First posted 2024-12-24 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Radiation Therapy; Gynecologic Cancer; Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Participants will either be randomized to the Immediate Start Group or to the Delayed Start Group.
  Participants in the:
  * Immediate Start Group: Sessions with the exercise coach will start during the first week of participants' radiation therapy, concurrently with radiation treatment and continue post-radiation.
  * Delayed Start Group: Sessions with the exercise coach will start 6-8 weeks after participants have completed radiation and continue 16-19 weeks post-radiation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Start Group (Experimental): Participants in this group will start the intervention during the first week of radiation therapy and continue through and post-completion of radiation
  Interventions: Behavioral: Exercise Coaching
- Delayed Start Group (Experimental): Participants in this group will start 6-8 weeks post - radiation and continue 16-19 weeks post-radiation.
  Interventions: Behavioral: Exercise Coaching

INTERVENTIONS:
Behavioral: Exercise Coaching — An exercise coaching program tailored for women with Stage I-IVA endometrial cancer who have undergone total or modified radical hysterectomy with surgical staging. The intervention targets a total of 8 participants who are planned to complete pelvic external beam radiation therapy as part of their adjuvant treatment.

SUMMARY:
Research has shown that for women who are undergoing pelvic radiation therapy, fatigue is a common side effect. Fatigue that occurs during radiation therapy can make it harder to perform daily living activities. While there are studies that recommend exercise as a treatment for fatigue in cancer patients and survivors, there are currently no studies that focus on the role of exercise for women undergoing pelvic radiation therapy. The purpose of this study is to see if incorporating an activity coaching program is helpful in improving treatment-related fatigue for women undergoing pelvic radiation therapy for endometrial cancer.

DETAILED DESCRIPTION:
The exercise coaching program is a program in which Participants will have ten weekly check-ins with a certified exercise coach. During check-ins, Participants and the exercise coach will set weekly goals. Participants will try to incorporate activities that are easy and enjoyable for them. These visits can be scheduled at their convenience and choose whether these check-ins will be in-person, or virtually.

All Participants who agree to join this study will be asked to:

* Participate in a program with an exercise coach to set weekly goals for activity. The timing of when the program will start will be based on the group Participants are assigned to.
* Receive a Fitbit to track how active they are, their heart rate and how many steps they've have taken.
* Complete 4 surveys which will be given throughout the course of the study.
* Complete a short 6-minute walking test to see how their heart and lungs respond to exercise. This test will be completed 4 times throughout the study.
* Participate in an interview with the principal investigator at the end of the study for feedback on how the study can be improved.

The study team expects to enroll 16 patients in this study. Participants will either be placed in the Immediate Start Activity Coaching Program or the Delayed Start Activity Coaching Program. 8 patients will be assigned to the Immediate Start Group, and 8 will be assigned to the Delayed Start Group. Participants will spend about 6 months in this study.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Pathologic diagnosis of endometrial cancer (any histology, Stage I-IVA)
* Has undergone modified radical or radical hysterectomy
* Plan to receive adjuvant treatment with pelvic external beam radiation therapy at ISCI
* ECOG performance status of 0-1
* Patient has a computer, smart phone, or tablet virtual access to the web-based platform and email
* Able to read, understand and provide written informed consent
* Deemed appropriate for unmonitored exercise by treating physician based on the following evidence-based criteria (1)

  * Walk without any assistance or assistance device
  * Absence of significant cognitive impairment
  * Absence of high risk for falls
* Participant does not need to refrain from any activity

Exclusion Criteria:

* Unable to schedule and attend coaching visits
* Participation in a regular exercise program of ≥150 minutes of moderate intensity exercise a week at baseline
* Unable to perform the five-times stand test
* Medical comorbidities including:

  * Unstable angina
  * Uncontrolled dysrhythmias
  * Acute pulmonary embolus
  * Active pulmonary infection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 16 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of a Randomized Trial: Participant Adherence to Exercise Coaching Sessions | Enrollment to end of follow up, up to 24 months
  Participant adherence to coaching sessions will be defined as complete adherence when engaging in 10 of the 10 planned exercise coaching sessions and high adherence as engaging in at least 7 of the planned 10 exercise coach check-ins. Participant adherence will be considered feasible if 70% of participants adhere to the coaching sessions.

SECONDARY OUTCOMES:
Change in patient-reported fatigue | Enrollment to end of follow up, up to 24 months
  Measurement of changes in the level of fatigue as reported by patients, using a Functional Assessment of Chronic Illness Therapy (FACIT) - Fatigue. FACIT-F fatigue subscale consists of 13 items. Patients rate the intensity of their fatigue symptoms on a scale of 0 to 4 (0=not at all and 4=very much). Total FACIT-F fatigue subscale score ranges from 0 to 52 with higher scores less fatigue and lower scores more fatigue
Change in patient-reported bowel/urinary toxicity | Enrollment to end of follow up, up to 24 months
  Assessment of changes in the severity of bowel and urinary toxicity symptoms, as reported by patients, using Expanded Prostate Cancer Index Composite (EPIC) bowel and urinary short form assessments. The EPIC-15 is a short-form version that includes 15 items across two domains: Urinary Function and Bowel Habits. Each item in the EPIC-15 is scored on a Likert scale, and the scores are transformed to a 0-100 scale, with higher scores indicating better quality of life.
Change in patient-reported Quality of Life (QOL) | Enrollment to end of follow up, up to 24 months
  Measurement of changes in the quality of life based on patient-reported outcomes, using Patient-Reported Outcomes Measurement Information System (PROMIS-29) Profile v2.1. It includes 29 items that assess seven key areas: Physical Function, Anxiety, Depression, Fatigue, Sleep Disturbance, Ability to Participate in Social Roles/Activities and Pain Interference. Each question usually has five response options ranging in value from one to five. The scores are then converted to T-scores using a scoring table. Higher T-Scores for Physical Function indicate better physical functioning, Higher T-Scores for Anxiety and Depression indicate more severe symptoms. Higher T-Scores for Fatigue and Sleep Disturbance indicate more fatigue or sleep problems. Higher T-Scores in ability to participate in social roles/activities indicate better ability to participate in social roles and activities. Higher T-Scores for Pain Interference means more interference from pain in daily activities and intense pain
Change in patient-reported cognitive function | Enrollment to end of follow up, up to 24 months
  Evaluation of cognitive function changes reported by patients, measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Cognitive Function Short Form 4a. This form contains 4 items. Each item is scored on a Likert scale from 1 (Never) to 5 (Very often). Raw scores are converted to T-scores using a scoring table. Higher T-scores indicate better cognitive function.
Change in patient-reported sexual function and satisfaction | Enrollment to end of follow up, up to 24 months
  Changes in sexual function and satisfaction, as reported by patients, using a Patient-Reported Outcomes Measurement Information System (PROMIS) Brief Profile Sexual Function and Satisfaction. Each item is scored on a Likert scale, and then converted into a T-Score. Higher T-scores indicate better sexual function and satisfaction.
Change in patient-reported self-efficacy | Enrollment to end of follow up, up to 24 months
  Measurement of changes in patients' perceived self-efficacy, using Patient-Reported Outcomes Measurement Information System (PROMIS) Self-Efficacy for Chronic Conditions. Each item is scored on a Likert scale, and then converted into a T-Score. Higher T-scores indicate greater self-efficacy.
Change in distance walked during the 6-Minute Walk Test (6MWT) | Enrollment to end of follow up, up to 24 months
  Measurement of the change in distance walked by patients during the 6-Minute Walk Test, a standardized test used to assess physical function.

CONTACTS AND LOCATIONS:
Overall Officials: Avani Rao, MD, Principal Investigator — Inova Health Care Services
Locations (4):
- United States (4):
  - Inova Schar Cancer Institute - Alexandria, Alexandria, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Inova Schar Cancer Institute - Fair Oaks, Fairfax, Virginia
  - Inova Schar Cancer Institute - Loudoun, Leesburg, Virginia

IPD SHARING:
Plan to Share IPD: Yes

DOCUMENTS (2):
  • Study Protocol (2025-05-12): https://cdn.clinicaltrials.gov/large-docs/28/NCT06746428/Prot_000.pdf
  • Informed Consent Form (2025-05-12): https://cdn.clinicaltrials.gov/large-docs/28/NCT06746428/ICF_001.pdf